CLINICAL TRIAL: NCT07045038
Title: BLOOD FLOW RESTRICTED RESISTANCE EXERCISES VERSUS LOW LEVEL LASER ON CARDIAC FUNCTIONS IN PATIENTS WITH CHRONIC HEART FAILURE
Acronym: heart failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samira Shukrey Shaffik Eshak, teaching assisstent, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resis versus LLL heart failure
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure NYHA Class II

STUDY DESIGN:
Intervention Model Description: 3 group of Heart failure patients Study Group A (20 patients) will receive blood flow restricted resistance exercises in addition to medical treatment program and routine cardiac rehabilitation.
  Study Group B (20 patients) will receive low level laser in addition to medical treatment program and routine cardiac rehabilitation.
  Control Group C (20 patients) will receive medical treatment program and routine cardiac rehabilitation only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture LLLT (Experimental): This mode of therapy will be conducted for study group B as follows:
  A therapeutic unit (M6 MLS from ASA laser, Italy) with wavelength 905 nm, output 5-20 MW, laser beam spot size 0.785 cm2, energy density 91 J/cm2, energy delivered 28 J, and frequency 500HZ. Laser probe will be placed in intercostal space both anteriorly and posteriorly on chest wall.
  Each acupuncture point will be stimulated with a laser for 60 s, three weekly sessions over 12 successive weeks. Anterior chest wall acupuncture points are {LU1, LU2, CV17, (Ren17)}, posterior chest wall from a prone or setting position of the patient {UB13, (BL13), UB 17(BL17
  Interventions: Device: Acupuncture LLLT:
- Blood flow restricted resistance exercise (Experimental): The subject will warm up and cool down for at least five to seven minutes each, (before and after exercise).
  The patients will perform blood flow restricted resistance exercise (BFRRE) at 40-80% of 1RM with 50% limb occlusion pressure (LOP), while placing cuff on midthigh and perform four sets of bilateral knee extension exercise, each set consist of 15 repetitions with 30-60 second rest in between sets and relieve cuff pressure in rest period, three weekly sessions over 12 successive weeks
  Interventions: Other: Blood flow restricted resistance exercise:
- Medical treatment and routine cardiac rehabilitation (Experimental): All patients will enroll to maximum doses guideline medical treatment that include (Beta blockers-Aspocid- Ator-Concor-Tritace).
  Also all patients will adhere to routine cardiac rehabilitation:
  The patients will enroll in CR program for 12 weeks, three times per week for 12 week. Moderate-intensity treadmill exercise training achieving a target heart rate of 40-60% of HR reserve (calculated from pre-exercise symptom-limited treadmill exercise stress test by modified Bruce protocol). The duration of each session was 30- 45 minutes (5-10 minutes of treadmill warm up, followed by 20-30 minutes of aerobic continuous treadmill training and terminated by 5-10 minutes of cooling down). The patients will be monitor by continuous ECG monitoring, recording of blood pressure, and heart rate
  Interventions: Drug: Medical treatment

INTERVENTIONS:
Device: Acupuncture LLLT: — Acupuncture LLLT:
  This mode of therapy will be conducted for study group B as follows:
  A therapeutic unit (M6 MLS from ASA laser, Italy) with wavelength 905 nm, output 5-20 MW, laser beam spot size 0.785 cm2, energy density 91 J/cm2, energy delivered 28 J, and frequency 500HZ. Laser probe will be placed in intercostal space both anteriorly and posteriorly on chest wall.
  Each acupuncture point will be stimulated with a laser for 60 s, three weekly sessions over 12 successive weeks. Anterior chest wall acupuncture points are {LU1, LU2, CV17, (Ren17)}, posterior chest wall from a prone or setting position of the patient {UB13, (BL13), UB 17(BL17)}.
  Arms: Acupuncture LLLT
Other: Blood flow restricted resistance exercise: — The subject will warm up and cool down for at least five to seven minutes each, (before and after exercise).
  The patients will perform blood flow restricted resistance exercise (BFRRE) at 40-80% of 1RM with 50% limb occlusion pressure (LOP), while placing cuff on midthigh and perform four sets of bilateral knee extension exercise, each set consist of 15 repetitions with 30-60 second rest in between sets and relieve cuff pressure in rest period, three weekly sessions over 12 successive weeks
  Arms: Blood flow restricted resistance exercise
Drug: Medical treatment — All patients will enroll to maximum doses guideline medical treatment that include (Beta blockers-Aspocid- Ator-Concor-Tritace).
  Also all patients will adhere to routine cardiac rehabilitation:
  The patients will enroll in CR program for 12 weeks, three times per week for 12 week. Moderate-intensity treadmill exercise training achieving a target heart rate of 40-60% of HR reserve (calculated from pre-exercise symptom-limited treadmill exercise stress test by modified Bruce protocol). The duration of each session was 30- 45 minutes (5-10 minutes of treadmill warm up, followed by 20-30 minutes of aerobic continuous treadmill training and terminated by 5-10 minutes of cooling down
  Arms: Medical treatment and routine cardiac rehabilitation

SUMMARY:
This study is designed to compare between blood flow restricted resistance exercises and low level laser on cardiac functions in patients with chronic heart failure

DETAILED DESCRIPTION:
This study will be carried out on sixty male and female patients diagnosed with chronic heart failure. They will be recruited from El-Demerdash hospital, Ain Shams university, Cairo. Their ages will be ranged from (40-60) years old. The design of this study will be a randomized controlled trail (RCT).

The patients of this study will randomly assigned into three equal groups (n=20):

Study Group A (20 patients) will receive blood flow restricted resistance exercises in addition to medical treatment program and routine cardiac rehabilitation.

Study Group B (20 patients) will receive low level laser in addition to medical treatment program and routine cardiac rehabilitation.

Control Group C (20 patients) will receive medical treatment program and routine cardiac rehabilitation only.

The program of treatment for the three groups A ,B , and C will be applied once per day, three times per week for 12 consecutive weeks

ELIGIBILITY:
Inclusion Criteria:

* 1- Sixty male and female patients diagnosed with chronic heart failure since six months with LVEF<40%.

  2- They are functionally classified as class II according to New York Heart Association (NYHA).

  3-Their age will be ranged from 40 to 60 years old. 4-Their BMI will be ranged from 25 to 29.9 kg/m². 5- They will have good mentality

Exclusion Criteria:

* - Unstable coronary heart disease. 2- Severe valvular diseases. 3- Underlying pulmonary disease (aspiration pneumonia, chronic obstructive pulmonary disease, pneumothorax, etc.).

  4- Inability to ambulate owing to physical problems (paresis induced by cerebral stroke, spinal cord injury, amputation, severe pain, dyspnea, etc.).

  5-muskloskletal problems (e.g. severe osteoarthritis or ankylosing spondylitis).

  6-impaired cognitive function (vascular dementia, Alzheimer's dementia, other psychological disease, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
: speckle-tracking echocardiography - NO Blood analysis | 3 months
  Echocardiography: speckle-tracking echocardiography an advanced, non invasive imaging modality that allow accurate assessment of the global and regional function of both atrial and ventricular chambers based on interaction between myocardial tissue and ultrasound beam. It is possible to obtain the deformation of LV myocardium along longitudinal, circumferential, radial and rotational plane. As longitudinal strain (LS) represents the LV myocardial shortening along its longitudinal axis. Radial strain (RS) reflect radial myocardial deformation corresponding to systolic thickening and is defined by positive curve. Circumferential strain (CR) represents the myocardial shortening along the circumferential plane, normally curves are negative.
  NO Blood analysis:
  All blood samples will be collected by venipuncture and immediately will be analyzed with Nitric Oxide Assay Kit (Fluorometric). The Kit is used to measure NO concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided